CLINICAL TRIAL: NCT04745676
Title: A Telehealth Advance Care Planning Intervention for Older Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Acronym: SICG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCO20134
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient (Experimental): The SICG program consists of the Serious Illness Conversation Guide as well as training and system-level support for physicians to conduct ACP conversations.
  Interventions: Behavioral: Telehealth; Behavioral: Control
- Caregiver (Experimental): The SICG program consists of the Serious Illness Conversation Guide as well as training and system-level support for physicians to conduct ACP conversations.
  Interventions: Behavioral: Telehealth; Behavioral: Control
- Oncology and Palliative Provider (Experimental): The SICG program consists of the Serious Illness Conversation Guide as well as training and system-level support for physicians to conduct ACP conversations.
  Interventions: Behavioral: Telehealth; Behavioral: Control

INTERVENTIONS:
Behavioral: Telehealth — Telehealth ACP intervention advance care planning intervention
Behavioral: Control — For the control arm, no telehealth visit will be scheduled.

SUMMARY:
This is a pilot study to evaluate the usability and feasibility of a telehealth-delivered advance care planning intervention among 20 older patients with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
Older adults with AML and MDS are more likely to receive aggressive care and less likely to utilize hospice at the end-of-life. Advance care planning (ACP) intervention delivered through telehealth may improve patient-reported outcomes and end-of-life care in this population. This pilot study seeks to evaluate the usability and feasibility of a telehealth-delivered advance care planning intervention. We will adapt the Serious Illness Care Program.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Age ≥60 years (conventional definition of older age in AML/MDS)
* AML or MDS diagnosis
* Being managed in the outpatient settings
* Able to provide informed consent
* English-speaking

Exclusion Criteria: N/A

Inclusion Criteria for Caregivers

* Age ≥21 years
* Selected by patient when asked if there is a "family member, partner, friend, or caregiver with whom you discuss or who can be helpful in health-related matters"
* Able to provide informed consent
* English-speaking

Exclusion Criteria: N/A

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — Univ. of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete and final study protocol will be made publicly available through the University of Rochester Cancer Center Community Oncology Research Program Research Base Protocol and Data Sharing Committee. The full protocol and data will be made publicly available no later than the publication date of the study findings from the final dataset. The protocol will include a detailed description of the study population, hypotheses tested, measurement and assessment information, data definitions and codes, and the analysis plan utilized. We will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing. Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years from accrual of the first subject.

REFERENCES:
- [Derived] LoCastro M, Wang Y, Yu T, Mortaz-Hedjri S, Mendler J, Norton S, Bernacki R, Carroll T, Klepin H, Wedow L, Goonan S, Erdos H, Bagnato B, Liesveld J, Huselton E, Kluger B, Loh KP. Clinicians' Perspectives on the Telehealth Serious Illness Care Program for Older Adults With Myeloid Malignancies: Single-Arm Pilot Study. JMIR Form Res. 2024 Jun 27;8:e58503. doi: 10.2196/58503. PMID 38935428
- [Derived] LoCastro M, Mortaz-Hedjri S, Wang Y, Mendler JH, Norton S, Bernacki R, Carroll T, Klepin H, Liesveld J, Huselton E, Kluger B, Loh KP. Telehealth serious illness care program for older adults with hematologic malignancies: a single-arm pilot study. Blood Adv. 2023 Dec 26;7(24):7597-7607. doi: 10.1182/bloodadvances.2023011046. PMID 38088668
- [Derived] LoCastro M, Sanapala C, Mendler JH, Norton S, Bernacki R, Carroll T, Klepin HD, Watson E, Liesveld J, Huselton E, O'Dwyer K, Baran A, Flannery M, Kluger B, Loh KP. Adaptation of Serious Illness Care Program to be delivered via telehealth for older patients with hematologic malignancy. Blood Adv. 2023 May 9;7(9):1871-1884. doi: 10.1182/bloodadvances.2022008996. PMID 36521100

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient; Caregiver; Clinician: The SICG program consists of the Serious Illness Conversation Guide as well as training and system-level support for physicians to conduct ACP conversations.
  Telehealth: Telehealth ACP intervention, advance care planning intervention
  For the control group, no telehealth visits were scheduled.
Period: Overall Study
Arm/Group | Patient | Caregiver | Clinician
Started | 20 | 6 | 10
Completed | 19 | 6 | 10
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population consists of 20 patients, 6 caregivers, and 9 clinicians (1 clinician did not provide demographic data).
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient | Caregiver | Clinician | Total
Number analyzed (Participants) | 20 | 6 | 9 | 35
Age, Continuous [Mean (Standard Deviation); unit: years]
  Patient | 75 (5.9) | 64 (13.7) | 44 (11.7) | 65.1 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Patient: Female | 9 | 4 | 6 | 19
  Patient: Male | 11 | 2 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 20 patients were included in the population of the study.
  Participants
    Patient: Hispanic or Latino | 0 | 0 | 0 | 0
    Patient: Not Hispanic or Latino | 16 | 5 | 9 | 30
    Patient: Unknown or Not Reported | 4 | 1 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 20 patients were included in the population of the study.
  Participants
    Patient: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Patient: Asian | 0 | 0 | 1 | 1
    Patient: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Patient: Black or African American | 1 | 0 | 0 | 1
    Patient: White | 17 | 6 | 8 | 31
    Patient: More than one race | 0 | 0 | 0 | 0
    Patient: Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Retention Rate
Description: Percentage of patients, caregivers, and clinicians who consented to the study, ultimately completing all study components
Time Frame: 12 Weeks
Population: Retention rate was focused for the patient and caregiver populations.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 20 | 6 | 10
Participants | 19 | 6 | 10

2. Primary Outcome: Recruitment Rate
Description: Number of patients, caregivers, and clinicians who are approached and agree to enroll.
Time Frame: 12 Weeks
Population: There are 29 patients analyzed because that many were approached, then 21 consented. One patient consented but withdrew before the intervention was initiated, leaving 20 enrolled participants. There were 7 caregivers approached, but 1 caregiver withdrew due to medical reasons. All 10 clinicians approached consented.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 29 | 7 | 10
Participants | 21 | 6 | 10

3. Primary Outcome: Mean Usability of the Telehealth Advance Care Planning Intervention Using the Telehealth Usability Questionnaire (TUQ)
Description: Telehealth Usability Questionnaire (TUQ) - A questionnaire (22 questions scored from 1 to 7, a higher score indicates greater usability) assessing the usability of telehealth implementation across the population (for patients or caregivers), the mean of all questions is then calculated, range 1-7, with an average of greater than 5 considered usable.
Time Frame: 12 Weeks
Population: Usability was an optional assessment, and 3 patients opted not to complete the survey. Therefore, data was not collected. All caregivers answered the survey. The clinicians were not included in the population of this aim.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 17 | 6 | 0
score on a scale | 5.9 (0.9) | 5.9 (1.1) |

4. Secondary Outcome: Pre- and Post-Intervention Change of the Mean Score for the General Anxiety Disorder-7 (GAD-7)
Description: General Anxiety Disorder-7 (GAD-7): A 7-item screening tool for anxiety (range 0-21, higher score indicates greater anxiety symptoms)
Time Frame: 12 Weeks
Population: General Anxiety Disorder-7 was an optional assessment, and 3 patients opted not to complete the survey. Therefore, data was not collected. All caregivers completed the survey. The clinicians were not included in the population of this aim.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 17 | 6 | 0
score on a scale | 0.1 (2.2) | -2.8 (5.0) |

5. Secondary Outcome: Pre- and Post-Intervention Change of the Mean Score for the Patient Health Questionnaire-9 (PHQ-9)
Description: Patient Health Questionnaire-9 (PHQ-9): A 9-item valid and reliable screening tool depression in the general population (range 0-27, higher score indicates greater depressive symptoms).
Time Frame: 12 Weeks
Population: Patient Health Questionnaire-9 was an optional assessment, and 3 patients opted not to complete the survey. Therefore, data was not collected. All caregivers completed the survey. The clinicians were not included in the population of this aim.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 17 | 6 | 0
score on a scale | 0.4 (4.2) | -1.0 (3.0) |

6. Secondary Outcome: Pre- and Post-Intervention Change of the Mean Score for the Distress Thermometer
Description: Distress Thermometer: A self-reported tool to screen for symptoms of distress, using a 0-10 rating scale (higher score indicates greater distress level).
Time Frame: 12 Weeks
Population: Distress Thermometer was an optional assessment, and 3 patients opted not to complete the survey. Therefore, data was not collected. All caregivers completed the survey. The clinicians were not included in the population of this aim.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 17 | 6 | 0
score on a scale | 0.3 (2.4) | -1.3 (1.4) |

7. Secondary Outcome: Pre- and Post-Intervention Change of the Mean Score for the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu)
Description: Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu): Consists of 17 questions on the general module and 17 leukemia-specific questions, score ranges from 0-176, higher score indicates better quality of life).
Time Frame: 12 Weeks
Population: Functional Assessment of Cancer Therapy-Leukemia was an optional assessment, and 2 patients opted not to complete the survey. Therefore, data was not collected. The caregivers and clinicians were not included in the population of this aim.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 18 | 0 | 0
score on a scale | -3.3 (17.6) |  |

8. Secondary Outcome: Post-Intervention Mean Score for the Health Care Communication Questionnaire (HCCQ)
Description: Health Care Communication Questionnaire (HCCQ): A questionnaire assessing patients' satisfaction with patient-oncologist communication (12 items, range from 12-60), higher score indicates greater satisfaction with communication.
Time Frame: 12 weeks
Population: Health Care Communication Questionnaire was an optional assessment, and 2 participants opted not to complete the survey. Therefore, data was not collected. All caregivers completed the survey. The clinicians were not included in the population of this aim.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Caregiver | Clinician
Number analyzed (Participants) | 18 | 6 | 0
score on a scale | 18.3 (2.1) | 18.2 (2.9) |

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Patients; Caregivers; Clinicians: The SICG program consists of the Serious Illness Conversation Guide as well as training and system-level support for physicians to conduct ACP conversations.
  Telehealth: Telehealth ACP intervention advance care planning intervention
Arm/Group | Patients | Caregivers | Clinicians
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/6 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04745676/Prot_SAP_000.pdf